CLINICAL TRIAL: NCT05480488
Title: A Single-center, Open-label Study to Investigate the Effect of Single- and Multiple-dose Daridorexant on the Pharmacokinetics of Midazolam and Its Metabolite 1-hydroxymidazolam, and the Effect of Single-dose Daridorexant on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Male Subjects
Brief Title: A Study to Examine the Effect of Daridorexant on the Way the Body Absorbs, Distributes, and Gets Rid of Midazolam and Warfarin in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Idorsia Pharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: ID-078-126
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Healthy
MeSH Terms: interventions — Midazolam; Warfarin; daridorexant

STUDY DESIGN:
Intervention Model Description: This is a prospective, open-label, fixed-sequence Phase 1 study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- • A (midazolam & warfarin), B (daridorexant, midazolam, & warfarin), & C (daridorexant & midazolam) (Other): * Treatment A - midazolam and warfarin: In the morning of Day 1, subjects will receive a single oral dose of 2 mg midazolam concomitantly with a single oral dose of 25 mg warfarin under fasted conditions.
  * Treatment B - daridorexant, midazolam, and warfarin: Subjects will receive an o.d. oral dose of 50 mg daridorexant in the morning from Day 1 to Day 7 under fasted conditions. In addition, in the morning of Day 1, the oral administration of 50 mg daridorexant will be followed 1 h later by a single oral dose of 2 mg midazolam concomitantly with a single oral dose of 25 mg warfarin under fasted conditions.
  * Treatment C - daridorexant and midazolam: In the morning of Day 1, subjects will receive a single oral dose of 50 mg daridorexant followed 1 h later by a single oral dose of 2 mg midazolam under fasted conditions.
  Interventions: Drug: Midazolam; Drug: Warfarin; Drug: Daridorexant

INTERVENTIONS:
Drug: Midazolam — Subjects will receive a single oral dose of 2 mg midazolam (Treatment A, B, and C).
Drug: Warfarin — Subjects will receive a single oral dose of 25 mg warfarin (Treatment A and B).
Drug: Daridorexant — Subjects will receive an o.d. oral dose of 50 mg daridorexant from Day 1 to Day 7 of Treatment B and a single oral dose of 50 mg daridorexant on Day 1 of Treatment C.

SUMMARY:
A study to examine the effect of daridorexant on the way the body absorbs, distributes, and gets rid of midazolam and warfarin in healthy male subjects

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent in a language understandable to the subject prior to any study-mandated procedure.
* Healthy male subject aged between 18 and 45 years (inclusive) at Screening.

Exclusion Criteria:

* Known hypersensitivity to daridorexant, midazolam, warfarin, or treatments of the same class, or any of their excipients.
* Any history of hemorrhagic disease, whether or not hereditary.
* Any history of complications with bleeding after surgery or tooth extractions and/or frequent nasal, hemorrhoidal, or gingival bleeding.
* Activated partial thromboplastin time (aPTT) > 40 sec and/or international normalized ratio (INR) > 1.15 at Screening.
* Platelet count < 150 or >400 x 10^9/L at Screening.
* Clinically relevant findings on the physical examination at Screening.
* Clinically relevant abnormalities on 12-lead ECG, measured after 5 min in the supine position at Screening.
* Clinically relevant findings in clinical laboratory tests (hematology, coagulation, clinical chemistry) at Screening.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-10-06 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) of midazolam and its metabolite 1-OH midazolam | Blood samples for pharmacokinetic analyses of midazolam will be taken at various time points from Day 1 to 2 of Treatment Period A, from Day 1 to 2 of Treatment Period B, and from Day 1 to 2 of Treatment Period C (total duration: 6 days).
Cmax of S-warfarin | Blood samples for pharmacokinetic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days).
Time to reach Cmax (tmax) of midazolam and 1-OH midazolam | Blood samples for pharmacokinetic analyses of midazolam will be taken at various time points from Day 1 to 2 of Treatment Period A, from Day 1 to 2 of Treatment Period B, and from Day 1 to 2 of Treatment Period C (total duration: 6 days).
Tmax of S-warfarin | Blood samples for pharmacokinetic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days).
Area under the concentration-time curve (AUC) from zero to infinity (AUC0-∞) of midazolam and 1-OH midazolam | Blood samples for pharmacokinetic analyses of midazolam will be taken at various time points from Day 1 to 2 of Treatment Period A, from Day 1 to 2 of Treatment Period B, and from Day 1 to 2 of Treatment Period C (total duration: 6 days)
AUC0-∞ of S-warfarin | Blood samples for pharmacokinetic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days).
Terminal elimination half-life (t½) of midazolam and 1-OH midazolam | Blood samples for pharmacokinetic analyses of midazolam will be taken at various time points from Day 1 to 2 of Treatment Period A, from Day 1 to 2 of Treatment Period B, and from Day 1 to 2 of Treatment Period C (total duration: 6 days).
T½ of S-warfarin | Blood samples for pharmacokinetic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days).

SECONDARY OUTCOMES:
AUC0-144 for international normalized ratio (AUC INR) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)
The maximum effect on INR (INRmax) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)
Time to reach maximum effect of INR (t Emax) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)
AUC0-144 for Factor VII (AUC VII) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)
The maximum effect on Factor VII (VIImax) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)
Time to reach maximum effect of Factor VII (t Emax) | Blood samples for pharmacodynamic analyses of S-warfarin will be taken at various time points from Day 1 to 7 of Treatment Period A and from Day 1 to 7 of Treatment Period B (total duration: 14 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Idosia Pharmaceuticals Ltd
Locations (1):
- Nuvisan GmbH, Neu-Ulm, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zenklusen I, Dingemanse J, Reh C, Gehin M, Kaufmann P. Effect of Daridorexant on the Pharmacokinetics of Midazolam, and on the Pharmacokinetics and Pharmacodynamics of Warfarin in Healthy Male Subjects. Drugs R D. 2024 Mar;24(1):97-108. doi: 10.1007/s40268-024-00456-8. Epub 2024 Mar 13. PMID 38472696